CLINICAL TRIAL: NCT06062134
Title: Pericapsular Nerve Group Block: An Imaging Study for Determination of the Spread of the Injectate Using 3-D CT Scan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philippe Gauthier (Other)
Responsible Party: Sponsor-Investigator, Philippe Gauthier, Principal Investigator, Centre Hospitalier Universitaire de Liege
Organization: Centre Hospitalier Universitaire de Liege (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-146
Record Dates: First submitted 2023-08-05; First posted 2023-10-02 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Post Operative Pain; Mechanisms of Analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: All subjects enrolled in the study received the same interventional regional analgesia technique (the pericapsular nerve group block) as part of the standard multimodal analgesia protocol. The local anesthetic was mixed with a radiocontrast agent in order to evaluate the spread of the injectate by using CT scan imaging.
Masking Description: No masking was required for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pericapsular nerve group block group (Experimental): All subjects enrolled in the study received a pericapsular nerve group block using a local anesthetic mixed with a contrast agent. After injection, subjects were transferred to the CT scan to obtain a 3D reconstruction to determine the spread of the injectate.
  Interventions: Procedure: Pericapsular nerve group block; Drug: 18 mL ropivacaine 0.5% + 2 mL radiopaque contrast

INTERVENTIONS:
Procedure: Pericapsular nerve group block — Ultrasound-guided injection of local anesthetic mixed with contrast agent underneath the iliopsoas muscle, lateral to the iliopsoas tendon.
Drug: 18 mL ropivacaine 0.5% + 2 mL radiopaque contrast — 20 mL of injectate: 18 mL ropivacaine 0.5% + 2 mL radiopaque contrast (Iomeron 300: 61.24% w/v of iomeprol equivalent to 30% iodine or 300 mg iodine/mL)

SUMMARY:
Over the last 20 years, different interventional regional analgesia techniques have been proposed to treat pain after hip surgeries.

The most commonly used techniques are the fascia iliaca and femoral nerve blocks, resulting in reduced pain scores, opioid-sparing effects, and opioid-related adverse effects. However, these interventional analgesia techniques result in a motor block and muscle weakness of the quadriceps muscle, impeding early ambulation and rehabilitation.

Recently, the pericapsular nerve group (PENG) block has been proposed as an effective choice for analgesia after hip surgeries while sparing the motor function of the lower extremities. The aim of this technique is to inject local anesthetic to target the more distal sensory branches innervating the anterior aspect of the hip joint.

DETAILED DESCRIPTION:
Ten patients scheduled for hip surgery were included after Ethical Committee approval and informed consent were obtained.

Preoperatively, patients received an ultrasound-guided pericapsular nerve group block. The injections were performed preoperatively using a Canon US Applio 700 with a linear transducer (14 to 6 MHz), and a 21-gauge, 80 mm stimulating needle (SonoPlex Stim, Pajunk ® ️ GmbH, Germany). After confirmation of the correct needle tip position with 2 mL of sodium chloride 0.9%, 20 mL of injectate containing 18 mL ropivacaine 0.5% with 2 mL of radiopaque contrast (Iomeron 300: 61.24% w/v of Iomeprol equivalent to 30% iodine or 300 mg iodine/mL (Bracco UK Limited)) was injected.

After surgery, high-definition CT scans (Siemens) were obtained to determine the distribution patterns of the injectates.

ELIGIBILITY:
Inclusion Criteria:

1. an indication for PENG blocks for postoperative pain management
2. American Society of Anesthesiologists (ASA) physical status I or II
3. at least 18 years old, and able to understand the purpose and risks of the study

Exclusion Criteria:

1. pregnancy
2. body mass index above 35 kg/m2
3. hepatic or renal insufficiency
4. history of allergic or adverse reactions to local anesthetics or contrast agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Concentration of the local anesthetic reaching specific anatomical areas of interest around the hip joint | 2 hours
  Computed tomography images will be used as measurement tool

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gautier, Principal Investigator — Anesthesiologist
Locations (1):
- Clinique Ste Anne-St Remi, Brussels, Belgium

REFERENCES:
- [Derived] Balocco AL, Gautier N, Van Boxstael S, Lopez AM, Carella M, Corten K, Sala-Blanch X, Hadzic A, Gautier PE. Pericapsular nerve group block: a 3D CT scan imaging study to determine the spread of injectate. Reg Anesth Pain Med. 2025 Jul 4;50(7):588-591. doi: 10.1136/rapm-2024-105459. PMID 38925712